CLINICAL TRIAL: NCT06897696
Title: Effect of Dexmedetomidine and Total Intravenous Anesthesia on Endothelial Damage-Related Biomarkers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Firat University (Other)
Responsible Party: Principal Investigator, Gulsum Altuntas, Faculty Member, Firat University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: ETHICAL APPROVAL 31335
Record Dates: First submitted 2025-03-13; First posted 2025-03-27 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Endothelial Damage; Dexmedetomidine; Syndecan 1; Heparan Sulpahate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- propofol+remifentanil (Active Comparator): to maintain anesthesia and analgesia propofol 5-8 mg/kg/h and remifentanil 5-10 µg/kg/h will be administered to all patients
  Interventions: Drug: propofol+remifentanyl group
- dexmedetomidine+propofol+remifentanyl group (Active Comparator): The dexmedetomidine+TIVA group will receive a bolus of 0.8-1 µg/kg dexmedetomidine for 10 minutes followed by continuous dexmedetomidine infusion at a rate of 0.3-0.5 µg/kg/hour.
  Interventions: Drug: Dexmedetomidine+propofol+remifentanyl group

INTERVENTIONS:
Drug: Dexmedetomidine+propofol+remifentanyl group — The dexmedetomidine+TIVA group will receive a bolus of 0.8-1 µg/kg dexmedetomidine for 10 minutes followed by continuous dexmedetomidine infusion at a rate of 0.3-0.5 µg/kg/hour.
  Arms: dexmedetomidine+propofol+remifentanyl group
Drug: propofol+remifentanyl group — propofol 5-8 mg/kg/h and remifentanil 5-10 µg/kg/h will be administered to all patients
  Arms: propofol+remifentanil

SUMMARY:
This study aimed to evaluate whether dexmedetomidine has a protective effect on endothelial damage by measuring plasma syndecan1 and heparan sulphate levels in rhinoplasty patients who take propofol+remifentanyl infusion.

DETAILED DESCRIPTION:
Endothelial Glycocalyx (EG) is a carbohydrate-rich network covering the apical surface of endothelial cells. It consists of sulphated glycoproteins linked to sialic acids (heparan sulphate, dermatan sulphate), core proteoglycans (mainly syndecan-1) and unsulphated glycosaminoglycans (CD 44) directly attached to the cytoplasmic membrane of endothelial cells. The fragile nature of endothelial glycocalyx makes it highly susceptible to damage, especially in critical diseases such as septic shock and inflammation, ischaemia-reperfusion (IR) syndrome, oxidative stress and major trauma. Endothelial glycocalyx damage worsens the patient's clinical outcome, leading to capillary leakage, tissue oedema, immune system disorders, and thrombosis.

Despite the widespread use of transmission electron microscopy, fluorescence microscopy and intravital microscopy in experimental investigations, these methods are not applicable at the bedside. The second most widely used method to investigate endothelial glycocalyx is biochemical analysis of EG degradation products (e.g. syndecan-1, heparan sulphate, hyaluronan).

In surgical procedures, general anaesthesia is a pharmacological method used to control pain and consciousness. The agents administered in this process may be associated with both hypnotic and analgesic mechanisms acting on the central nervous system and side effects on the autonomic nervous system and circulatory system. Pharmacological agents used during general anaesthesia may exert pro-inflammatory or anti-inflammatory effects on the endothelium directly or indirectly. Some anaesthesia modalities may trigger endothelial damage by increasing oxidative stress, free radical production and the release of inflammatory cytokines. On the other hand, some techniques may show endothelial protective properties; this is related to the dose, duration and pharmacodynamic properties of the agents used. Because there is no pharmacological agent to prevent EG damage, it is important to prevent EG degradation in patients undergoing surgery. For all these reasons, evaluating the effects of general anaesthesia on endothelial function may provide important information for the protection of vascular health during and after surgery.

This study aimed to evaluate whether dexmedetomidine has a protective effect on endothelial damage in rhinoplasty patients under general anaesthesia by measuring plasma syndecan1 and heparan sulphate levels.

ELIGIBILITY:
Inclusion Criteria:patients between the ages of 18-50 who will undergo rhinoplasty will be included in the study -

Exclusion Criteria:patients who do not agree to participate in the study, patients with underlying peripheral arterial disease, coronary artery disease, hypertension, diabetes mellitus, and ASA (American Society of Anaesthesiologists) Classification ≥3 will be excluded.

-

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2025-04-10 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
endothelial damage in patients under general anaesthesia | from preoperative 24 hours to postoperative 24 hours
  The relationship between increased serum Syndecan-1 and Heparan Sulfate levels and endothelial damage in patients under general anaesthesia

SECONDARY OUTCOMES:
dexmedetomidine protection against endothelial damage | from preoperative 24 hours to postoperative 24 hours
  Difference in endothelial damage between the patients receiving dexmedetomidine and those not receiving dexmedetomidine

CONTACTS AND LOCATIONS:
Overall Officials: Gulsum Altuntas, Study Chair — Firat University
Locations (1):
- Firat University Hospital, Elâzığ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
study protocol will be shared with other researchers
Supporting Information: Study Protocol
Time Frame: from 2025 december
Access Criteria: all researchers